CLINICAL TRIAL: NCT00713726
Title: Post-Operatory Analgesia in Newborn Infants: a Comparative Study of Fentanyl Versus Tramadol
Brief Title: Tramadol Versus Fentanyl for Post-Operative Analgesia in Newborn Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Albert B. Sabin Vaccine Institute (Other)
Responsible Party: Ruth Guinsburg, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1386/06
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2008-07

CONDITIONS: Pain; Neonatal Infections; Analgesia
Keywords: Pain; Analgesia; Newborn Infant; Opioids; Side-effects; Intensive care; Postoperative
MeSH Terms: conditions — Pain; Agnosia | interventions — Fentanyl; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- F (Active Comparator): Patients that received continued infusion of fentanyl at a steady dose for the first 48 hours and, then, doses were gradually decreases until stop
  Interventions: Drug: FentanyL
- T (Experimental): Patients that received continued infusion of tramadol at a steady dose for the first 48 hours and, then, doses were gradually decreases until stop
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: FentanyL — Fentanyl: 1 µg/kg/h for preterm infants and 2 µg/kg/h for term infants for 48 hours and than gradually decrease until interruption of the drug.
  Arms: F
Drug: Tramadol — Tramadol: 0.1 mg/kg/h for preterm infants and 0.2 mg/kg/h for term infants for 48 hours and than gradually decrease until interruption of the drug.
  Arms: T

SUMMARY:
In newborn infants submitted to surgical procedures, tramadol may provide an effective analgesia and decrease the time on mechanical ventilation support and the time to achieve full enteral feeding.

ELIGIBILITY:
Inclusion Criteria:

* Infant 0-28 days of life with indication of large or medium surgical procedure (definition according to the American College of Cardiology, American Heart Association - 2002)

Exclusion Criteria:

* Death or hospital discharge until 72 hours after surgical procedure
* New surgery until 72 hours after the studied surgical procedure
* Proved bacterial infection before surgery
* Ambiguous genitalia
* Chromosomal syndromes

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Pain assessment wuth CRIES and NFCS pain scales during the first 72 hours after surgical procedure | Every 2-4h during the first 72 hours after surgical procedure

SECONDARY OUTCOMES:
Time between surgical procedure and successful extubation | Hospital stay
Time between surgical procedure and achievement of 100 mL/kg of enteral feeding | hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Guinsburg, MD, Study Director — Federal University of São Paulo; Ana Julia C Alencar, Principal Investigator — Federal university of são Paulo and Albert Sabin Hospital
Locations (1):
- Albert Sabin Hospital, Fortaleza, Ceará, Brazil

REFERENCES:
- [Derived] Alencar AJ, Sanudo A, Sampaio VM, Gois RP, Benevides FA, Guinsburg R. Efficacy of tramadol versus fentanyl for postoperative analgesia in neonates. Arch Dis Child Fetal Neonatal Ed. 2012 Jan;97(1):F24-9. doi: 10.1136/adc.2010.203851. Epub 2011 Apr 5. PMID 21471025